CLINICAL TRIAL: NCT03776058
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Safety, Tolerability, and Clinical Effects of Twice-daily Doses of an Oral Calcimimetic Agent (AMG 073) in Subjects With Primary Hyperparathyroidism (HPT)
Brief Title: Safety, Tolerability, and Clinical Effects of Twice-daily Doses of Cinacalcet (AMG 073) in Adults With Primary Hyperparathyroidism (HPT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00990160
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cinacalcet (Experimental): Participants received 65 mg cinacalcet orally twice a day for 4 weeks.
  Interventions: Drug: Cinacalcet
- Placebo (Placebo Comparator): Participants received placebo to cinacalcet orally twice a day for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinacalcet — Tablets for oral administration
  Other Names: AMG 073; Sensipar®; Mimpara®
  Arms: Cinacalcet
Drug: Placebo — Tablets for oral administration
  Arms: Placebo

SUMMARY:
The primary objectives were to assess the safety and tolerability of twice daily (BID) doses of 65 mg cinacalcet administered orally to adults with primary HPT.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years old before beginning of screening
* Use, in the opinion of the principal investigator, effective contraceptive measures throughout the study
* Negative serum pregnancy test within 15 days before day 0
* Plasma iPTH concentration > 45 pg/mL on at least 2 occasions (during the screening phase) at least 7 days apart
* Serum calcium concentration ≥ 11 mg/dL on 2 occasions (during the screening phase) at least 7 days apart
* Acceptable renal function, with an estimated creatinine clearance > 50 mL/min as determined by the Cockroft and Gault equation
* Acceptable hepatic function, defined as serum aspartate transaminase (AST), alanine transaminase (ALT), and total bilirubin ≤ 2 times the upper limit of normal (central laboratory's range)
* Laboratory test results within the central laboratory's normal range for hematology, coagulation, urinalysis, and clinical chemistry parameters not mentioned specifically in other inclusion/exclusion criteria
* Chest x-ray within the past 12 months, with no evidence of an active infectious, inflammatory, or malignant process
* Informed consent for participation in the study

Exclusion Criteria:

* Any unstable medical condition requiring hospitalization within 30 days before day 0, or otherwise unstable condition in the judgment of the investigator
* Awaiting or scheduled for parathyroidectomy within 2 months after study day 0
* Pregnant or nursing
* Received, within 21 days before day 0, therapy with systemic glucocorticoids (> 5 mg/day prednisone or equivalent), lithium, tricyclic antidepressants (with the exception of amitriptyline and nortriptyline), thioridazine, haloperidol, flecainide, drugs with a narrow therapeutic index that are primarily metabolized by hepatic cytochrome P450 CYP 2D6, drugs that affect renal tubular calcium handling (ie, thiazide or loop diuretics), or calcitonin
* Dose changes in bisphosphonates, thyroid replacement therapy, selective estrogen receptor modulators (SERMs), or changes in daily doses of estrogen (greater than 0.75 mg) within 90 days before day 0
* Subjects who discontinued estrogen or SERM therapy must have been off treatment for at least 90 days before day 0.
* Alcohol or illicit drug abuse within 12 months before day 0 based on self-report
* Myocardial infarction within 6 months before day 0
* Ventricular rhythm disturbance requiring current treatment
* Seizure within 12 months before day 0
* History (within 5 years) of malignancy of any type, other than nonmelanomatous skin cancers or in situ cervical cancer
* Evidence (within 5 years) of treatment for and/or active sarcoidosis, tuberculosis, or diseases other than primary HPT known to cause hypercalcemia
* History of familial hypocalciuric hypercalcemia (FHH)
* Uncontrolled diabetes, as defined by hemoglobin A1c (HbA1c) ≥ 8.0
* Gastrointestinal disorder that may be associated with impaired absorption of orally administered medications
* Inability to swallow tablets similar in size to an aspirin tablet
* Known sensitivity to products administered during the study
* Previous participation as a subject in this study (ie, withdrawn early) or a prior study involving AMG 073 administration
* Enrolled in, or not yet completed at least 28 days since ending other investigational device or drug trial(s)
* Psychiatric disorder that would interfere with understanding and giving informed consent or compliance with protocol requirements
* Any other condition that might reduce the chance of obtaining data (ie, known poor compliance) required by the protocol or that might compromise the ability to give truly informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2000-06-15 (Actual); Primary Completion 2000-12-26 (Actual); Study Completion 2000-12-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 4 weeks
Number of Participants with Clinically Significant Laboratory Tests, Vital Signs or Electrocardiogram Assessments | 4 weeks

SECONDARY OUTCOMES:
Percent Change from Baseline in Serum Calcium | Baseline and week 4
Percent Change from Baseline in Plasma Intact Parathyroid Hormone (iPTH) | Baseline and week 4
Percent Change from Baseline in Bone-specific Alkaline Phosphatase (BALP) | Baseline and week 4
Percent Change from Baseline in 1,25 dihydroxy Vitamin D3 | Baseline and week 4
Percent Change from Baseline in Serum Phosphorus | Baseline and week 4
Percent Change from Baseline in N-telopeptide (NTx) | Baseline and week 4
Percent Change from Baseline in Urine Osmolality | Baseline and week 4
Percent Change from Baseline in Calcium/Creatinine Ratio | Baseline and week 4
Percent Change from Baseline in Phosphorus/Creatinine Ratio | Baseline and week 4
Percent Change from Baseline in N-telopeptide/Creatinine Ratio | Baseline and week 4